CLINICAL TRIAL: NCT03978468
Title: Interagency Collaboration To Improve Home Care of Children With Medical Complexity.
Brief Title: ICOLLAB FOR Children With Medical Complexity
Acronym: ICOLLAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00058144; 10359 (Other Grant/Funding Number: Health Resources and Services Administration)
Record Dates: First submitted 2019-06-05; First posted 2019-06-07 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2022-06

CONDITIONS: Children With Medical Complexity
Keywords: Collaboration, Home Health Nurse, Providers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Group (Active Comparator): Children will receive usual care.
  Interventions: Other: Usual Care
- Interagency Collaboration (ICollab Group) (Experimental): Subjects of this arm will receive ICollab intervention in addition to usual care which consists of communication with Home Health Nurse (HHN) , Collaborative meetings, and communication with Primary Care Physician (PCP)
  Interventions: Other: Interagency Collaboration (ICollab); Other: Usual Care

INTERVENTIONS:
Other: Interagency Collaboration (ICollab) — The intervention has the following components: 1) ICollab Component 1: The Nurse Clinician will review clinic and emergency room (ER) visit notes for clinicians' recommendations and communicate these to the home health nurse (HHN). 2) ICollab Component 2a: The intervention team will meet weekly by phone with HHNs (6 times/ child). The Nurse Clinician will document meeting notes for each child in the ER, communicate this information with the HHN, and share it with the primary care provider (PCP) by routing the note through the ER or faxing the note. 3) ICollab Component 2b: The Nurse Clinician will be available as a resource for the HHN during regular work hours for clinical problem-solving. 4) ICollab Component 2c: the intervention team physician will offer her contact information for clinical problem-solving about the child to the PCP. The Nurse Clinician will communicate with the PCP about the plan developed in the meetings, and changes to plan of care.
  Arms: Interagency Collaboration (ICollab Group)
Other: Usual Care — The primary medical team identifies the need for home health nursing services for Children with Medical Complexity(CMC), and the hospital care coordinators help caregivers choose a home health agency. Hospital-based physicians write home health orders that are communicated to the home health agency. The clinic manager of the home health agency uses these orders to develop the home health plan of care, Centers for Medicare & Medicaid Services(Form CMS-485) and communicates the plan to the agencies' HHNs. PCPs oversee the home health plan of care.

SUMMARY:
Background: Children with medical complexity (CMC) have higher hospitalizations and readmissions compared to children without medical complexity. While CMC were institutionalized in the past, increasingly CMCs are now cared for at home. Caring for individuals with disabilities at home, and not congregate care settings is a Healthy People 2020 Objective. Home health nursing, especially good-quality care, is important for CMC. The purpose of this research is to test whether collaboration between home health nurses, primary-care doctors, and the complex care team (a special team at Brenner Children's Hospital that provides care for children with complex chronic medical conditions (CCMC)) can improve the health of these children.

DETAILED DESCRIPTION:
The specific aims of this study are to: develop and implement a model of care, Interagency Collaboration (ICollab) in which communication with Home Health Nurse (HHN) and Primary Care Provider (PCP) is maintained and clinical support is provided to HHN; evaluate whether ICollab is effective in reducing healthcare utilization of Children with medical complexity (CMC) and caregiver burden; and assess caregiver satisfaction in home health care, HHN retention, and collaboration with other healthcare providers.

Methods: Investigators will develop and implement an intervention model (ICollab) that includes: (1) maintaining communication with HHN and PCP about clinical information about CMC, and (2) providing clinical support to HHN. Investigators will create an interdisciplinary intervention team in our children s hospital consisting of a pediatrician and a nurse. The intervention team will ensure communication with HHN and PCP by communicating clinical information (recommendations from clinic visits and emergency room (ER) visits, and discharge summary). The team will provide clinical support to HHN via collaborative meetings and availability as a resource for clinical problem-solving with HHN. Investigators will recruit 110 CMC discharged home on private-duty nursing services into this randomized trial. The intervention group (n=55) will receive the ICollab intervention for 6 months post-discharge from the hospital, in addition to usual care. Children in the control group (n=55) will receive only usual care. Outcome measures will include healthcare utilization metrics (hospitalization rates, ER visit rates, and days to readmission), caregiver burden and caregiver satisfaction with home health care, HHN retention, and HHN collaboration with other healthcare providers. Investigators hypothesize that ICollab will reduce healthcare utilization and caregiver burden, and improve caregiver satisfaction with home health care, increase HHN retention, and increase HHN collaboration with other healthcare providers. Investigators will perform a systematic process evaluation of the implementation of the intervention and standardize the ICollab model.

Implications: How healthcare delivery of CMC can be structured to avoid fragmentation especially surrounding transition across clinical settings is an understudied area. Our results will address this gap by providing a critically needed evidence-base for interventions to improve the quality of healthcare delivery for CMC

ELIGIBILITY:
Inclusion Criteria:

* The Nurse Clinician will screen children for eligibility for the study (see Eligibility Form). Only children with medical complexity (CMC) who are discharged home with private-duty nursing (PDN) services will be included. CMC will be identified as (1) child <18 years of age; and (2) presence of a chronic condition, defined as a health condition expected to last ≥ 12 months; and (3) complexity of the condition, defined as needing ongoing care with ≥ 5 sub-specialists/ services, or dependent on ≥ 2 technologies (e.g. gastrostomy, oxygen, tracheostomy, ventilator, etc.).

Exclusion Criteria:

* Children who might turn 18 during the intervention period will be excluded to avoid having to re-consent with adult informed consent form (ICF). Children who receive skilled nursing visits or personal care services only, those discharged to a long-term care facility or to a foster home, or whose caregivers do not speak English/Spanish, will be excluded.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2019-11-08 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Rate of Hospitalization | 6 months
  Using data obtained from the Translational Data Warehouse, the number of hospitalizations will be calculated for each child..compare the rate of hospitalizations/ 100-child years in the 2 groups. Number of hospitalizations during the observation period will be counted and the rate will be calculated as:
  [Number of hospitalizations/ observation period in years] *100
Rate of ER visits | 6 months
  Rate of ER visits will be calculated as follows: [Number of ER visits/ observation period in years]*100
Days to readmission | 6 months
  Days to readmission will be calculated as the duration between the time of index hospitalization (time of enrollment) and the date of admission for the subsequent hospitalization.

SECONDARY OUTCOMES:
Impact on Family Scale | 6 months
  Change in caregiver burden will be measured using the 15- item Impact on Family Scale - Revised, which has 4 domains - financial, family/ social, personal strain, and mastery. Scores range from 15 to 60; the lower the score, the greater the impact.
Client Satisfaction Survey | 6 months
  Caregiver satisfaction with home care will be compared between the 2 groups and measured by the Client Satisfaction Survey. It has 35 items with 4 subscales. Total Score: Minimum 1 and Maximum 5; lower the score the better

OTHER OUTCOMES:
Home health nurse retention | 6 months
  Staff retention will be measured as turnover rate using data from monthly caregiver surveys. [Average monthly HHN separations/average number of HHN assigned to the case] *100
Home health nurse-healthcare provider collaborations, HHN PCP ICOLLAB Survey | 6 months
  Caregiver perception of collaboration between HHN and other healthcare providers at the end of the study period will be compared for the 2 groups. HHN PCP ICOLLAB Survey. Qualitative data analysis methods will be used

CONTACTS AND LOCATIONS:
Overall Officials: Savithri Nageswaran, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nageswaran S, Easterling D, Ingram CW, Skaar JE, Miller-Fitzwater A, Ip EH. Randomized controlled trial evaluating a collaborative model of care for transitioning children with medical complexity from hospital to home healthcare: Study protocol. Contemp Clin Trials Commun. 2020 Dec;20:100652. doi: 10.1016/j.conctc.2020.100652. Epub 2020 Sep 18. PMID 32964166

DOCUMENTS (1):
  • Informed Consent Form (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/68/NCT03978468/ICF_000.pdf